CLINICAL TRIAL: NCT03030131
Title: A Phase II Prospective Immune Neoadjuvant Therapy Study od Durvalumab (MEDI4736) in Early Stage Non-small Cell Lung Cancer
Brief Title: Immune Neoadjuvant Therapy Study of Durvalumab in Early Stage Non-small Cell Lung Cancer
Acronym: IONESCO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Definitive discontinuation according to safety monitoring of death from the 46th patient onwards.
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-1601
Record Dates: First submitted 2017-01-12; First posted 2017-01-24 (Estimated); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: IFCT; neodjuvant; immune therapy; Non small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab (Experimental): durvalumab 750 mg IV J1, J15, J29
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — durvalumab 750 mg IV Day1, 15, 29
  Other Names: MEDI4736

SUMMARY:
Lung cancer is still the leading cause of cancer related-deaths worldwide, with an overall all-stage 5-year survival of approximately 17%. The primary treatment of early stage (I-IIIA) NSCLC is curative surgery. Although patients treated with curative surgery have a better prognosis, the 5-year survival for patients treated with surgery alone remains low, ranging from 67% (stage IA) to 23% (stage IIIA). Several randomized trials comparing postoperative chemotherapy versus no chemotherapy have shown a significant overall survival benefit from postoperative chemotherapy in completely resected patients with NSCLC stage II and IIIA. Likewise other randomized trials have demonstrated preoperative chemotherapy improves survival and recently the analyses also based on individual patients data of 15 randomized trials showed a significant benefit of preoperative chemotherapy on survival with the same survival improvement of 5% at 5 years. Then, neoadjuvant chemotherapy has also become accepted in many countries.

Targeting of PD-1 receptors and its ligand PD-L1, and inhibiting their engagement is an attractive therapeutic option in the early stage NSCLC, which may reactivate host immune responses and enable longterm tumor control.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of primary non-small cell carcinoma of the lung.
* Tissue block of diagnosis must be available for submission after inclusion (one HES slide and one paraffin embedded block).
* Patients must be classified clinically as Stage IB (only T = 4 cm in greatest dimension, N0), Stage IIA (T2b,N0) and some of Stage IIB : (T1-2,N1) and (T3 : > 5 cm and ≤ 7 cm in greatest dimension surrounded by lung or associated with separate tumor nodule(s) in the same lobe but without mediastinum or chest wall involvements, or superior sulcus tumors, N0) on the basis of clinical evaluation (8th classification TNM, UICC 2015). In case of invasion of the main bronchus (distance < 2 cm from carina), a biopsy of the carina is required. A pre-surgical PET scan of the thorax and a MRI or CT scan of the brain as well as thorax abdomen pelvis CT scan must be done prior to surgery and before inclusion. If preoperative CT and/or PET are suspicious for mediastinal nodal involvement, invasive mediastinal staging with mediastinoscopy or EBUS-TBNA must be performed. Station 5 or 6 lymph nodes may be accessed by anterior mediastinotomy or VATS.
* Pre-operative (neo-adjuvant) platinum based or other chemotherapy except the treatment of the protocol is not permissible. Pre-operative radiation therapy is not permissible
* The patient must have an ECOG performance status of 0, 1.
* Hematology (done within 14 days prior to inclusion and with values within the ranges specified below): If anemic, patients should be asymptomatic and should not be decompensated. Transfusions are permissible.

Haemoglobin ≥ 9,0 g/dL Absolute neutrophil count > 1.5 x 109/L or > 1,500/µl Platelets > 100 x 109/L or > 100,000/µl

- Biochemistry (done within 14 days prior to inclusion and with values within the ranges specified below): Total bilirubin* within normal institutional limits Alkaline phosphatase < 2.5 x institutional upper limit of normal AST(SGOT) and ALT(SGPT) < 2.5 x institutional upper limit of normal Creatinine Clearance > 40 ml/min TSH within normal institutional limits

* excluding Gilbert's syndrome

Creatinine clearance to be measured directly by 24 hour urine sampling or as calculated by Cockcroft Formula:

Females: GFR = 1.04 x (140-age) x weight in kg serum creatinine in μmol/L Males: GFR = 1.23 x (140-age) x weight in kg serum creatinine in μmol/L

* Other investigations detailed in Section 6 must have been performed within the timelines indicated.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to inclusion in the trial to document their willingness to participate.
* Patients must be accessible for treatment and follow-up. Investigators must assure themselves the patients included on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.
* Protocol treatment is to begin within 7 days of patient inclusion
* Age of at least 18 years.
* Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: ≥60 years old and no menses for ≥ 1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
* Females of childbearing potential who are sexually active with a nonsterilized male partner or men who are sexually active with women of childbearing potential must use a highly effective method of contraception prior the first dose of investigational product, and must agree to continue using such precautions for 4 months after the final dose of investigational product. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception.

Exclusion Criteria:

* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer, or other solid tumours curatively treated with no evidence of disease for > 5 years following the end of treatment and which, in the opinion of the treating physician, do not have a substantial risk of recurrence of the prior malignancy.
* A combination of small cell and non-small cell lung cancer or pulmonary carcinoid tumour.
* History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. NOTE: patients with Grave's disease and/or psoriasis not requiring systemic therapy within the last two years from inclusion are not excluded.
* History of primary immunodeficiency, history of allogenic organ transplant, use of immunosuppressive agents within 28 days of inclusion* or a prior history of severe (grade 3 or 4) immune mediated toxicity from other immune therapy.

  * NOTE: Intranasal/inhaled corticosteroids or systemic steroids that do not to exceed 10 mg/day of prednisone or equivalent dose of an alternative corticosteroid are permissible.
* Live attenuated vaccination administered within 30 days prior to inclusion.
* History of hypersensitivity to durvalumab or any excipient.
* Patients who have experienced untreated and/or uncontrolled cardiovascular conditions and/or have symptomatic cardiac dysfunction (unstable angina, congestive heart failure, myocardial infarction within the previous year or cardiac ventricular arrhythmias requiring medication, history of 2nd or 3rd degree atrioventricular conduction defects). Patients with a significant cardiac history, even if controlled, should have a LVEF > 50% within 12 weeks prior to inclusion.
* Concurrent treatment with other investigational drugs or anti-cancer therapy.
* Patients with active or uncontrolled infections or with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol. This includes but is not limited to:

  * known prior history of tuberculosis;
  * known acute hepatitis B or C by serological evaluation;
  * known Human immunodeficiency virus infection.
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
* Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* Known history of previous clinical diagnosis of tuberculosis
* Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Surgical resection R0 | 2 months
  Patient percentage of surgical resection R0 after a maximum of 3 cycles of immune therapy

SECONDARY OUTCOMES:
Response Rate (recist 1.1) | After 28 days (3 cycles of immune therapy maximum)
Metabolic response rate on TEP-FDG | After 28 days (3 cycles of immune therapy maximum)
Delay between surgery and start of treatment | After 28 days (3 cycles of immune therapy maximum)
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 month
Disease-Free Survival (DFS) | 1 year
  Time from the date of inclusion to the date of first documented disease relapse or the occurrence of a new invasive primary malignancy or death from any cause
Overall survival (OS) | 1 year
  Time from the inclusion to the date of death of any cause, or censored at their last known alive date
Evaluation of predictive/prognostic value of PD-1/PD-L1 expression | 1 month
Evaluation of changes in plasma/serum cytokines and other biomarkers | 1 month
Major Pathological Response | 2 months

CONTACTS AND LOCATIONS:
Locations (31):
- France (31):
  - Amiens - Clinique de l'Europe, Amiens
  - Argenteuil - CH, Argenteuil
  - Bayonne - CH, Bayonne
  - Bordeaux - Institut Bergonié, Bordeaux
  - Caen - CHU, Caen
  - Caen - CRLCC, Caen
  - Chauny - CH, Chauny
  - Clermont-Ferrand - CHU, Clermont-Ferrand
  - Cornebarrieu - Clinique des Cèdres, Cornebarrieu
  - Grenoble - CHU, Grenoble
  - Le Mans - CHG, Le Mans
  - Limoges - CHU, Limoges
  - Mantes La Jolie - CH, Mantes-la-Jolie
  - AP-HM Hopital Nord, Marseille
  - Marseille - Hôpital Européen, Marseille
  - Metz - Hôpital Robert Schuman, Metz
  - Mulhouse - CH, Mulhouse
  - Nancy - Polyclinique Gentilly, Nancy
  - Nantes - CRLCC, Nantes
  - Paris - Hopital Tenon, Paris
  - Paris - HEGP, Paris
  - Paris - Hôpital Cochin, Paris
  - Paris - Montsouris, Paris
  - Paris - Saint Joseph, Paris
  - Paris Bichat, Paris
  - Pau - CHG, Pau
  - Centre René Huguenin, Saint-Cloud
  - Institut de Cancérologie de l'Ouest - site René Gauducheau, Saint-Herblain
  - Saint-Quentin - CH, Saint-Quentin
  - Strasbourg - NHC, Strasbourg
  - Toulouse - CHU Larrey, Toulouse

REFERENCES:
- [Derived] Wislez M, Mazieres J, Lavole A, Zalcman G, Carre O, Egenod T, Caliandro R, Dubos-Arvis C, Jeannin G, Molinier O, Massiani MA, Langlais A, Morin F, Le Pimpec Barthes F, Brouchet L, Assouad J, Milleron B, Damotte D, Antoine M, Westeel V. Neoadjuvant durvalumab for resectable non-small-cell lung cancer (NSCLC): results from a multicenter study (IFCT-1601 IONESCO). J Immunother Cancer. 2022 Oct;10(10):e005636. doi: 10.1136/jitc-2022-005636. PMID 36270733
- See also: Site web — http://www.ifct.fr/index.php/fr/la-recherche/item/2041-ifct-1601-ionesco

DOCUMENTS (1):
  • Study Protocol (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT03030131/Prot_000.pdf